CLINICAL TRIAL: NCT06911229
Title: Neurophysiology of Locomotor Adaptation and Freezing of Gait in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB202401786; R21AG088600 (NIH)
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
Keywords: Freezing of gait; deep brain stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DBS ON (Active Comparator): DBS will be turned on
  Interventions: Device: Deep Brain Stimulation (DBS)
- DBS OFF (No Intervention): DBS will be turned off

INTERVENTIONS:
Device: Deep Brain Stimulation (DBS) — Patients will receive DBS in the clinically-optimized setting.
  Arms: DBS ON

SUMMARY:
Locomotor adaptation will be studied using an established split-belt treadmill paradigm, consisting of baseline (1:1 speed ratio), split-belt adaptation (2:1) and post-adaptation (1:1) walking. Split-belt walking will be performed under DBS ON and DBS OFF conditions, while off-medication.

DETAILED DESCRIPTION:
We will test the hypotheses that DBS can facilitate split-belt walking adaptation with DBS ON compared with DBS OFF.

ELIGIBILITY:
Inclusion Criteria:

* consensus diagnosis of idiopathic PD by fellowship trained movement disorders neurologists at the Normal Fixel Institute of Neurological Diseases;
* chronically stable DBS, defined as having had DBS for at least 6 months in duration with optimized DBS settings;
* Age between 18 - 80 years old per the FDA data sheet for PD DBS;
* no dementia according to the clinical diagnostic criteria for PD dementia;
* ambulatory without the use of walking aids, or another person's assistance.

Exclusion Criteria:

* other previous neurological surgery;
* suspicion of other neurologic diagnoses such as atypical parkinsonism, or Alzheimer's disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Step length rate of adaptation | 1 hour
  The rate of adaptation in step length asymmetry is estimated by fitting an exponential decay function to step length asymmetry over the first 100 strides in adaptation.
Step length magnitude of adaptation | 1 hour
  The magnitude of adaptation in step length asymmetry is estimated by fitting an exponential decay function to step length asymmetry over the first 100 strides in adaptation.
Step length after-effects | 1 hour
  The after-effect in step length asymmetry is calculated as the mean difference in step length asymmetry between the last 5 strides of baseline and the first 5 series of post-adaptation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States